CLINICAL TRIAL: NCT07100405
Title: A Prospective, Non-interventional Study of TACE Combined With PD-1 Inhibitor in Patients With Advanced Hepatocellular Carcinoma: Efficacy and Immune Microenvironment Dynamics
Brief Title: TACE Combined With Anti-PD-1 Antibody in Patients With Advanced Hepatocellular Carcinoma: Study on Efficacy and Immune Microenvironment
Acronym: TASK-01-RW
Status: Recruiting | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Peng Wang, professor, Fudan University
Other Study IDs: TASK-01-RW
Record Dates: First submitted 2025-07-27; First posted 2025-08-03 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A baseline tumor biopsy and blood collection before initiation of treatment, followed by a second tumor biopsy with paired blood collection after the first response evaluation will be planned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TACE+PD1 inhibitor
  Interventions: Drug: PD-1 inhibitor; Procedure: TACE

INTERVENTIONS:
Drug: PD-1 inhibitor — An approved agent (e.g., Pembrolizumab, Nivolumab, Sintilimab, Tislelizumab, etc.) will be selected based on clinical practice and administered at standard doses and schedules.
Procedure: TACE — TACE is performed by using embolic agent combined with Lipiodol-pirarubicin emulsion per Investigator decision

SUMMARY:
This is a prospective, non-interventional, observational study evaluating the efficacy and immune microenvironment changes in Patients with Advanced Hepatocellular Carcinoma treated with TACE Combined with PD-1 Inhibitor.

DETAILED DESCRIPTION:
This is a prospective, non-interventional, observational study evaluating the efficacy and immune microenvironment changes in Patients with Advanced Hepatocellular Carcinoma treated with TACE Combined with PD-1 Inhibitor. The primary endpoint is objective response rate (ORR), with secondary endpoints including disease control rate (DCR), duration of response (DOR), time to response (TTR), progression-free survival (PFS), overall survival (OS), and immune profiling of tumor tissue and peripheral blood before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* BCLC stage C, and stage B who are not amenable to curative or locoregional therapies.
* Diagnosis of hepatocellular carcinoma.
* At least one measurable site of disease as defined by modified RECIST (mRECIST) criteria with spiral CT scan or MRI.
* No prior anticancer therapy, including TACE/HAIC, chemotherapy, targeted therapy, or immunotherapy).
* Planned to receive TACE plus anti-PD1 inhibitor as first-line treatment.
* ECOG performance status 0-1.
* Adequate organ function:
* ANC ≥1.5 × 10⁹/L, platelets ≥60 × 10⁹/L, hemoglobin ≥9 g/dL.
* Total bilirubin ≤1.5 × ULN, AST/ALT ≤3 × ULN (≤5 × ULN if liver metastases).
* Creatinine ≤1.5 × ULN or CrCl ≥60 mL/min.
* Willing to provide archival/fresh tumor tissue and peripheral blood samples.
* Signed informed consent.

Exclusion Criteria:

* Prior systemic therapy.
* Active autoimmune disease requiring immunosuppression.
* Active infection requiring IV antibiotics.
* HIV-positive or active HBV/HCV infection (HBsAg+ with HBV DNA ≥2000 IU/mL; HCV RNA+).
* Symptomatic CNS metastases.
* Pregnancy/lactation.
* Any condition compromising protocol compliance or data interpretation per investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a prospective, non-interventional, observational study evaluating the efficacy and immune microenvironment changes in Patients with Advanced Hepatocellular Carcinoma treated with TACE Combined with PD-1 Inhibitor.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) evaluated by the investigator per Response Evaluation Criteria in Solid Tumors Version 1.1 | max 24 months
  ORR is defined as the percentage of participants who have a confirmed complete response (CR: disappearance of all target lesions) or partial response (PR: at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters). Responses are according to RECIST 1.1 as assessed by investigator.

SECONDARY OUTCOMES:
Disease control rate (DCR) evaluated by the investigator per Response Evaluation Criteria in Solid Tumors Version 1.1 | max 24 months
  DCR is defined as the proportion of patients with complete response (CR), partial response (PR) and stable disease (S.D)
Duration of Response (DOR) evaluated by the investigator per Response Evaluation Criteria in Solid Tumors Version 1.1 | max 24 months
  DOR is defined as the time from first documented complete or partial response until disease progression, death from any cause, or censoring at date of last tumor assessment.
Time to Response (TTR) evaluated by the investigator per Response Evaluation Criteria in Solid Tumors Version 1.1 | max 24 months
  TTR is defined as the time from the start of treatment until the first objective observation of a response (either partial response, PR, or complete response, CR), provided that the response is subsequently confirmed
Progression Free Survival (PFS) evaluated by the investigator per Response Evaluation Criteria in Solid Tumors Version 1.1 | max 24 months
  PFS is defined as the time from study treatment to disease progression or all-cause death as assessed by the investigator (whichever occurs first)
Overall survival (OS) evaluated by the investigator per Response Evaluation Criteria in Solid Tumors Version 1.1 | max 42 months
  OS is defined as the time from study treatment to the date of death of the subject, regardless of the cause of death
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | max 42 months
  An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The percentage of participants who experience at least one AE will be reported.

OTHER OUTCOMES:
Translational study | max 42 months
  Proportion of different immune cell types in tumors based on single-cell RNA sequencing between two groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No